CLINICAL TRIAL: NCT01347710
Title: A Phase 3, Open Label, Multicenter Study for the Assessment of Myocardial Perfusion Using Positron Emission Tomography (PET) Imaging of Flurpiridaz F18 Injection in Patients With Suspected or Known Coronary Artery Disease (CAD)
Brief Title: A Phase 3 Multi-center Study to Assess PET Imaging of Flurpiridaz F 18 Injection in Patients With CAD.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BMS747158-301
Record Dates: First submitted 2011-04-11; First posted 2011-05-04 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2014-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease.; Positron Emission Tomography Myocardial Perfusion Imaging.; Single Positron Emission Computed Tomography.; Flurpiridaz F18 Injection.
MeSH Terms: conditions — Coronary Artery Disease | interventions — BMS 747158-02; Technetium Tc 99m Sestamibi; technetium tc-99m tetrofosmin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flurpiridaz F18 (Experimental): Open-label study of a single dose of Flurpiridaz F18 injection for PET MPI compared to a single dose of 99mTc sestamibi or tetrofosmin for SPECT MPI in patients with suspected or known coronary artery disease referred for coronary catheterization
  Interventions: Drug: Flurpiridaz F18; Drug: 99mTechnicium (sestamibi or tetrofosmin)

INTERVENTIONS:
Drug: Flurpiridaz F18 — Injection of Flurpiridaz F18 for the purposes of PET myocardial profusion imaging (MPI) analysis
  Other Names: flurpiridaz F 18
Drug: 99mTechnicium (sestamibi or tetrofosmin) — Injection of 99mTc sestamibi or tetrofosmin for the purposes of SPECT MPI analysis
  Other Names: 99mTc sestamibi or 99mTc Tetrofosmin

SUMMARY:
The primary objective of the study is to assess the diagnostic efficacy (specificity and sensitivity) of flurpiridaz F18 injection PET myocardial perfusion imaging (MPI) compared to single photon emission computed tomography (SPECT) MPI in the detection of significant coronary artery disease (CAD) as defined by invasive coronary angiography (ICA) or a documented history of Myocardial Infarction (MI).

DETAILED DESCRIPTION:
The study will assess the diagnostic efficacy (sensitivity and specificity) of Flurpiridaz F18 Injection MPI against SPECT MPI in patients screened for CAD as determined by ICA. Six hundred and eighty evaluable patients will be enrolled and will undergo SPECT MPI and Flurpiridaz F18 PET MPI. Patients will be considered for enrollment if they are scheduled to undergo or have undergone prior ICA without intervention (being either positive or negative for CAD).

ELIGIBILITY:
Inclusion Criteria:

Invasive Coronary Angiography. Men or Women age 18 or older - see protocol for additional details.

Exclusion Criteria:

Women who are pregnant, lactating, or of child bearing potential who are not practicing birth control.

Unstable cardiac status. History of coronary artery bypass graft. History of percutaneous coronary intervention within the past six months. See protocol for additional details.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 795 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Orlandi, MD, Study Director — Lantheus Medical Imaging
Locations (81):
- United States (73):
  - Cardiology Associates of Mobile, Inc., Mobile, Alabama
  - Scottsdale Medical Imaging, Ltd., Scottsdale, Arizona
  - West Side Medical Associates of Los Angeles, Beverly Hills, California
  - USC PET Imaging Science Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - VA West Los Angeles Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Veterans Affairs Palo Alto Health Care System, Palo Alto, California
  - Cardiovascular Consultants Medical Group, Pleasant Hill, California
  - Northern California PET Imaging Center-Palo Alto, Sacramento, California
  - VA San Diego Healthcare System, San Diego, California
  - UCSF Medical Center, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Alfieri Cardiology, Newark, Delaware
  - Christiana Care Health System, Newark, Delaware
  - Elite Research and Clinical Trials, Aventura, Florida
  - Independent Imaging, LLC, Boynton Beach, Florida
  - Coastal Cardiology Consultants dba The Heart & Vascular Institute of Florida, Clearwater, Florida
  - Florida Heart Associates, Fort Myers, Florida
  - St. Luke's Cardiology Associates, Jacksonville, Florida
  - The Cardiovascular Center, PA, Lake Mary, Florida
  - Florida Hospital/Cardiovascular Institute (Florida Heart Group), Orlando, Florida
  - South Florida Research Solutions, Pembroke Pines, Florida
  - Memorial Hospital of Tampa, Tampa, Florida
  - Georgia Health Sciences Univ/Med College of GA, Augusta, Georgia
  - South Coast Imaging Center, Savannah, Georgia
  - Gateway Cardiology, PC, Jerseyville, Illinois
  - Norton Cardiovascular Associates, Louisville, Kentucky
  - Biomedical Research Foundation of Northwest Louisiana, Shreveport, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Mass General Hospital (MGH), Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State University - Harper University Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. Mary's Healthcare (Trinity Health), Grand Rapids, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Missouri Cardiovascular Specialists, LLP, Columbia, Missouri
  - Cardiovascular Imaging Technologies (CVIT), Kansas City, Missouri
  - Saint Louis University School of Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Las Vegas Radiology, Las Vegas, Nevada
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Pinnacle Health Cardiovascular Institute/ Associated Cardiologists, Harrisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Presbyterian University Hospital, Pittsburgh, Pennsylvania
  - Berks Cardiologists, Ltd., Wyomissing, Pennsylvania
  - York Hospital /Wellspan Health, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Center for Biomedical Research, Knoxville, Tennessee
  - Cardiovascular Research of Knoxville - St. Mary's Health Care System, Inc., Knoxville, Tennessee
  - Vanderbilt Heart and Vascular Institute, Nashville, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Excel Diagnostics and Nuclear Oncology Center, Houston, Texas
  - Katy Cardiology, Katy, Texas
  - West Houston Area Clinical Trial Consultants, LLC, Tomball, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - McGuire Veteran Affairs Medical Center, Richmond, Virginia
  - Carilion Cardiology Clinic, Roanoke, Virginia
  - Roanoke Heart Institute, Roanoke, Virginia
- Canada (4):
  - University of Western Ontario, London, Ontario
  - KMH Cardiology and Diagnostic and MRI Centres, Mississauga, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turku PET Centre, Turku
- Puerto Rico (2):
  - San Patricio MEDFLIX (San Patricio MRI & CT Center), Guaynabo
  - VA Caribbean Healthcare System, San Juan

REFERENCES:
- [Derived] Lopez DM, Huck DM, Divakaran S, Brown JM, Weber BN, Lemley M, Builoff V, Shanbhag A, Lan Z, Buckley C, Al-Mallah MH, Dorbala S, Blankstein R, Slomka P, Di Carli MF. Utility of 18F-Flurpiridaz PET Relative Flow Reserve in Differentiating Obstructive From Nonobstructive Coronary Artery Disease. Circ Cardiovasc Imaging. 2025 Nov;18(11):e018323. doi: 10.1161/CIRCIMAGING.125.018323. Epub 2025 Oct 9. PMID 41064867
- [Derived] Poitrasson-Riviere A, Moody JB, Renaud JM, Hagio T, Arida-Moody L, Buckley CJ, Al-Mallah MH, Nallamothu BK, Weinberg RL, Ficaro EP, Murthy VL. Integrated myocardial flow reserve (iMFR) assessment: optimized PET blood flow quantification for diagnosis of coronary artery disease. Eur J Nucl Med Mol Imaging. 2023 Dec;51(1):136-146. doi: 10.1007/s00259-023-06455-2. Epub 2023 Oct 9. PMID 37807004
- [Derived] Hagio T, Moody JB, Poitrasson-Riviere A, Renaud JM, Pierce L, Buckley C, Ficaro EP, Murthy VL. Multi-center, multi-vendor validation of deep learning-based attenuation correction in SPECT MPI: data from the international flurpiridaz-301 trial. Eur J Nucl Med Mol Imaging. 2023 Mar;50(4):1028-1033. doi: 10.1007/s00259-022-06045-8. Epub 2022 Nov 19. PMID 36401636
- [Derived] Maddahi J, Lazewatsky J, Udelson JE, Berman DS, Beanlands RSB, Heller GV, Bateman TM, Knuuti J, Orlandi C. Phase-III Clinical Trial of Fluorine-18 Flurpiridaz Positron Emission Tomography for Evaluation of Coronary Artery Disease. J Am Coll Cardiol. 2020 Jul 28;76(4):391-401. doi: 10.1016/j.jacc.2020.05.063. PMID 32703509

RESULTS

PARTICIPANT FLOW:
Groups:
- Flurpiridaz F 18: Open-label study of a single dose of Flurpiridaz F18 injection for PET MPI compared to SPECT MPI in patients with suspected or known coronary artery disease referred for coronary catheterization
Period: Overall Study
Arm/Group | Flurpiridaz F 18
Started | 795
Completed | 764
Not Completed | 31
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 4
Not completed — Angio or SPECT not completed | 18
Not completed — issue with vitals prior to dosing | 1
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: Safety population, received at least one dose of flurpiridaz F 18
Arm/Group | Flurpiridaz F 18
Number analyzed (Participants) | 795
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 458
  >=65 years | 337
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249
  Male | 546
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43
  Not Hispanic or Latino | 708
  Unknown or Not Reported | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 105
  White | 652
  More than one race | 0
  Unknown or Not Reported | 24

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Efficacy of Flurpiridaz F 18 PET Myocardial Perfusion Imaging (MPI) Sensitivity Versus SPECT Myocardial Perfusion Imaging Sensitivity
Description: Diagnostic efficacy of one day rest and stress flurpiridaz F 18 PET MPI sensitivity versus SPECT MPI sensitivity in the detection of coronary artery disease (CAD) by majority rule using invasive coronary angiography as the truth standard,
Time Frame: 60 days
Population: All safety evaluable patients who had rest and stress flurpiridaz F 18 PET MPI and SPECT MPI procedures resulting in evaluable data, and had evaluable invasive coronary angiography
Measure: Number (95% Confidence Interval); unit: Proportion of true positive cases
Groups:
- Flurpiridaz F18 PET MPI: Open-label study of a single dose of Flurpiridaz F18 injection for PET MPI compared to SPECT MPI in patients with suspected or known coronary artery disease referred for coronary catheterization
  Flurpiridaz F18: Injection of Flurpiridaz F18 for the purposes of PET MPI analysis
Arm/Group | Flurpiridaz F18 PET MPI
Number analyzed (Participants) | 755
Proportion of true positive cases
  PET MPI sensitivity | .719 [.670 to .763]
  SPECT MPI Sensitivity | .537 [.485 to .588]
Statistical Analysis 1: Comparison: Flurpiridaz F18 PET MPI; Test type: Superiority or Other; p < 0.001, McNemar — P-value for sensitivity comparison of flurpiridaz F18 PET MPI vs SPECT MPI for majority rule; Two-sided McNemar's (chi-squared) test superiority

2. Secondary Outcome: Diagnostic Efficacy of Flurpiridaz F18 PET MPI Sensitivity Versus SPECT MPI Sensitivity in Subgroups: Pharmacologic Stress, Females and BMI>/=30.
Description: Diagnostic efficacy of flurpiridaz F18 PET MPI sensitivity versus SPECT MPI sensitivity by majority rule in the detection of CAD using invasive coronary angiography as the truth standard, , in subgroups: pharmacologic stress, females and BMI >/=30. Value reported is the number of true positives, i.e. True Positive: Patients with abnormal MPI and disease positive by the truth standard
  I
Time Frame: 60 days
Population: all safety evaluable patients who had a rest and stress flurpiridaz F18 PET MPI and SPECT MPI procedures resulting in evaluable data and evaluable invasive coronary angiography
Measure: Number (95% Confidence Interval); unit: proportion of true postives
Groups:
- Flurpiridaz F18 PET MPI: Open-label study of a single dose Flurpiridaz F18 injection for PET MPI compared to SPECT MPI in patients with suspected or known coronary artery disease referred for coronary catheterization
  Flurpiridaz F18: Injection of Flurpiridaz F18 for the purposes of PET MPI analysis
Arm/Group | Flurpiridaz F18 PET MPI
Number analyzed (Participants) | 755
proportion of true postives
  PET sensitivity pharmacologic stress | 0.736 [.679 to .785]
  SPECT sensitivity pharmacologic stress | 0.533 [.472 to .592]
  PET sensitivity in females | 0.644 [.517 to .754]
  SPECT sensitivity in females | 0.356 [.246 to .483]
  PET sensitivity BMI >/=30 | 0.722 [.653 to .782]
  SPECT sensitivity BMI >/=30 | 0.533 [.461 to .605]
Statistical Analysis 1: Comparison: Flurpiridaz F18 PET MPI; Test type: Superiority or Other; p < 0.001, McNemar — p-Value for sensitivity comparison of flurpiridaz F18 PET MPI vs SPECT MPI for majority rule in patients under going pharmacologic stress; Two-sided McNemar's (chi-squared) test superiority
Statistical Analysis 2: Comparison: Flurpiridaz F18 PET MPI; Test type: Superiority or Other; p < 0.001, McNemar — p-Value for sensitivity comparison of flurpiridaz F18 PET MPI vs. SPECT MPI for majority rule in females; p-Value based on two-sided McNemar's (Chi-squared) test superiority
Statistical Analysis 3: Comparison: Flurpiridaz F18 PET MPI; Test type: Superiority or Other; p < 0.001, McNemar — p-Value for sensitivity comparison of flurpiridaz F18 PET MPI vs SPECT MPI for majority rule in patients with BMI >/=30; p-Value based on two-sided McNemar's (Chi-squared) test superiority

3. Secondary Outcome: Diagnostic Efficacy of Flurpiridaz F18 PET MPI Specificity Versus SPECT Specificity in Subgroups: Pharmacologic Stress, Females and BMI>/=30.
Description: Diagnostic efficacy of flurpiridaz F18 PET MPI specificity versus SPECT specificity by majority rule in the detection of CAD using invasive coronary angiography as the truth standard, in subgroups: pharmacologic stress, females and BMI >/=30. Value represents the number of true negative, i.e. True Negative: Patients with normal MPI and disease negative by the truth standard
Time Frame: 60 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of true negatives
Arm/Group | Flurpiridaz F18 PET MPI
Number analyzed (Participants) | 755
proportion of true negatives
  PET MPI specificity pharmacological stress | .773 [.720 to .819]
  SPECT MPI specificity pharmacological stress | .875 [.831 to .909]
  PET MPI specificity females | .795 [.730 to .848]
  SPECT MPI specificity females | .869 [.812 to .911]
  PET MPI specificity BMI >/=30 | .777 [.719 to .826]
  SPECT MPI specificity BMI >/=30 | .850 [.798 to .89]
Statistical Analysis 1: Comparison: Flurpiridaz F18 PET MPI; Test type: Non-Inferiority or Equivalence — Systematic review of literature and meta-analysis of diagnostic efficacy of SPECT MPI to evaluate the performance criteria of SPECT MPI in studies with various levels of control. Analysis of study BMS747158-201. Non-inferiority margin (delta) = 7%; p = 0.891, Z test — p-Value for specificity comparison of flurpiridaz F18 PET MPI vs. SPECT MPI for majority rule in patients undergoing pharmacologic stress; z test for non inferiority for specificity
Statistical Analysis 2: Comparison: Flurpiridaz F18 PET MPI; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = .546, z test — p-Value for specificity comparison of flurpiridaz F18 PET MPI vs. SPECT MPI for majority rule in female patients; z test for non-inferiority for specificity
Statistical Analysis 3: Comparison: Flurpiridaz F18 PET MPI; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = .538, z test — p-Value for specificity comparison of flurpiridaz F18 PET MPI vs. SPECT MPI for majority rule BMI >/=30; z test for non-inferiority for specificity

4. Secondary Outcome: Diagnostic Performance Evaluation of Localization of CAD for Sensitivity (PETVsSPECT).
Description: Overall sensitivity of flurpiridaz F18 PET MPI in coronary territories (Qualitative Diagnosis vs. SPECT MPI by majority rule vs. truth standard (angiographic stenosis greater than or equal to 50% stenosis and confirmed MI); left descending coronary artery (LAD), left circumflex artery (LCX), right coronary artery (RCA), and non - LAD. Value reported is the number of true positives, i.e. True Positive: Patients with abnormal MPI and disease positive by the truth standard
Time Frame: 60 days
Population: All safety evaluable patients who had rest and stress flurpiridaz F 18 Flurpiridaz F18 PET MPI and SPECT MPI procedures resulting in evaluable data, and had evaluable invasive coronary angiography
Measure: Number (95% Confidence Interval); unit: Proportion of true positives
Groups:
- Flurpiridaz F 18: Open-label study of a single dose Flurpiridaz F18 injection for PET MPI compared to SPECT MPI in patients with suspected or known coronary artery disease referred for coronary catheterization
Arm/Group | Flurpiridaz F 18
Number analyzed (Participants) | 755
Proportion of true positives
  PET sensitivity LAD | .495 [.430 to .561]
  SPECT sensitivity LAD | .333 [.275 to .398]
  PET sensitivity LCX | .398 [.331 to .469]
  SPECT sensitivity LCX | .251 [.195 to .317]
  PET sensitivity RCA | .596 [.528 to .661]
  SPECT sensitivity RCA | .476 [.409 to .544]
  PET sensitivity Non-LAD | .627 [.568 to .682]
  SPECT sensitivity Non-LAD | .464 [.406 to .523]
Statistical Analysis 1: Comparison: Flurpiridaz F 18; Test type: Superiority or Other; p < 0.001, McNemar — p-Value for sensitivity comparison of flurpiridaz F18 PET MPI and SPECT MPI for majority rule in the localization of coronary artery disease; LAD; Two-sided McNemar (chi-squared) test superiority for sensitivity; LAD
Statistical Analysis 2: Comparison: Flurpiridaz F 18; Test type: Superiority or Other; p < 0.001, McNemar — p-Value for sensitivity comparison of flurpiridaz F18 PET MPI and SPECT MPI for majority rule in the localization of coronary artery disease; LCX; p-Value based on two-sided McNemar's (Chi-squared) test superiority for sensitivity; LCX
Statistical Analysis 3: Comparison: Flurpiridaz F 18; Test type: Superiority or Other; p < 0.001, McNemar — p-Value for sensitivity comparison of flurpiridaz F18 PET MPI and SPECT MPI for majority rule in the localization of coronary artery disease; RCA; p-Value based on two-sided McNemar's (Chi-squared) test superiority for sensitivity; RCA
Statistical Analysis 4: Comparison: Flurpiridaz F 18; Test type: Superiority or Other; p < 0.001, McNemar — p-Value for sensitivity comparison of flurpiridaz F18 PET MPI and SPECT MPI for majority rule in the localization of coronary artery disease; Non-LAD; p-Value based on two-sided McNemar's (Chi-squared) test superiority for sensitivity; Non-LAD

5. Secondary Outcome: Diagnostic Performance Evaluation of Localization of CAD for Specificity (PETVsSPECT).
Description: Overall specificity of flurpiridaz F18 PET MPI in Coronary Territories (Qualitative Diagnosis) vs. SPECT MPI by majority rule vs. truth standard (angiographic stenosis greater than or equal to 50% stenosis and confirmed MI); left descending coronary artery (LAD), left circumflex artery (LCX), right coronary artery (RCA), and non - LAD. Value represents the number of true negative, i.e. True Negative: Patients with normal MPI and disease negative by the truth standard
Time Frame: 60 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of true negatives
Arm/Group | Flurpiridaz F 18
Number analyzed (Participants) | 755
proportion of true negatives
  PET specificity LAD | .867 [.835 to .893]
  SPECT specificity LAD | .932 [.908 to .951]
  PET specificity LCX | .904 [.877 to .926]
  SPECT specificity LCX | .970 [.952 to .981]
  PET specificity RCA | .845 [.812 to .873]
  SPECT specificity RCA | .912 [.886 to .933]
  PET specificity Non-LAD | .814 [.777 to .846]
  SPECT specificity Non-LAD | .923 [.895 to .943]
Statistical Analysis 1: Comparison: Flurpiridaz F 18; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = .379, z Test — p-Value for specificity comparison of flurpiridaz F18 PET MPI and SPECT MPI for majority rule in the localization of coronary artery disease; LAD; z test for non-inferiority for specificity; LAD
Statistical Analysis 2: Comparison: Flurpiridaz F 18; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = .358, Z Test — p-Value for specificity comparison of flurpiridaz F18 PET MPI and SPECT MPI for majority rule in the localization of coronary artery disease; LCX; z test for non-inferiority for specificity; LCX
Statistical Analysis 3: Comparison: Flurpiridaz F 18; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = .442, z Test — p-Value for specificity comparison of flurpiridaz F18 PET MPI and SPECT MPI for majority rule in the localization of coronary artery disease; RCA; z test for non-inferiority for specificity; RCA
Statistical Analysis 4: Comparison: Flurpiridaz F 18; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = .984, z Test — p-Value for specificity comparison of flurpiridaz F18 PET MPI and SPECT MPI for majority rule in the localization of coronary artery disease; Non-LAD; z test for non-inferiority for specificity; non-LAD

6. Secondary Outcome: Diagnositic Performance Evaluation of Multivessel Disease (PETvsSPECT).
Description: Overall summary of sensitivity for identifying multi-vessel disease between flurpiridaz F18 PET MPI and SPECT MPI by majority rule vs. truth standard (angio >/=50% stenosis and confirmed MI). Value reported is the number of true positives, i.e. True Positive: Patients with abnormal MPI and disease positive by the truth standard
Time Frame: 60 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of true positives
Arm/Group | Flurpiridaz F18 PET MPI
Number analyzed (Participants) | 755
proportion of true positives
  PET MPI sensitivity; multivessel disease | .410 [.340 to .484]
  SPECT MPI sensitivity; multivessel disease | .275 [.215 to .345]
Statistical Analysis 1: Comparison: Flurpiridaz F18 PET MPI; Test type: Superiority or Other; p < 0.001, McNemar — p-Value of sensitivity for flurpiridaz F18 PET MPI vs. SPECT MPI for majority rule; multivessel disease; p-Value based on two-sided McNemar's (Chi squared) test superiority

7. Secondary Outcome: Diagnositic Performance Evaluation of Multivessel Disease (PETvsSPECT).
Description: Overall summary of specificity for identifying multi-vessel disease between flurpiridaz F18 PET MPI and SPECT MPI by majority rule vs. majority rule (angio >/=50% stenosis and confirmed MI). Value represents the number of true negative, i.e. True Negative: Patients with normal MPI and disease negative by the truth standard
Time Frame: 60 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of true negatives
Arm/Group | Flurpiridaz F18 PET MPI
Number analyzed (Participants) | 755
proportion of true negatives
  PET MPI specificity; multivessel disease | .882 [.853 to .906]
  SPECT MPI specificity; multivessel disease | .964 [.945 to .976]
Statistical Analysis 1: Comparison: Flurpiridaz F18 PET MPI; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.827, z test — p-Value of specificity for comparison of flurpiridaz F18 PET MPI vs. SPECT MPI in detecting multivessel disease; p-Value based on one-sided z test for non-inferiority

8. Secondary Outcome: Overall Summary of Sensitivity of PET MPI vs SPECT MPI; Image Quality Excellent or Good
Description: Overall summary of sensitivity of flurpiridaz F18 PET MPI (qualitative image quality of excellent or good) vs. SPECT MPI by majority rule vs. truth standard(angio >/=50% stenosis and confirmed MI). Value reported is the number of true positives, i.e. True Positive: Patients with abnormal MPI and disease positive by the truth standard
Time Frame: 60 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of true positives
Arm/Group | Flurpiridaz F18 PET MPI
Number analyzed (Participants) | 755
proportion of true positives
  PET MPI sensitivity; image quality excellent/good | .711 [.658 to .759]
  SPECT MPI sensitivity image quality excellent/good | .539 [.483 to .594]
Statistical Analysis 1: Comparison: Flurpiridaz F18 PET MPI; Test type: Superiority or Other; p < 0.001, McNemar — p-Value for sensitivity comparison of flurpiridaz F18 PET MPI vs SPECT MPI for majority rule; image quality of excellent or good; p-Value based on two-sided McNemar's (Chi-squared) test superiority for sensitivity

9. Primary Outcome: Diagnostic Efficacy of Flurpiridaz PET MPI Specificity Versus SPECT MPI Specificity
Description: Diagnostic efficacy of flurpiridaz PET MPI specificity versus SPECT MPI specificity by majority rule in the detection of CAD using invasive coronary angiography as the truth standard
Time Frame: 60 days
Population: all safety evaluable patients who had rest and stress flurpiridaz F 18 PET MPI and SPECT MPI procedures resulting in evaluable data and had evaluable invasive coronary angiography
Measure: Number (95% Confidence Interval); unit: Proportion of true negatives
Groups:
- Flurpiridaz F18: Open-label study of a single dose of Flurpiridaz F18 injection for PET MPI compared to SPECT MPI in patients with suspected or known coronary artery disease referred for coronary catheterization
  Flurpiridaz F18: Injection of Flurpiridaz F18 for the purposes of PET MPI analysis
Arm/Group | Flurpiridaz F18
Number analyzed (Participants) | 755
Proportion of true negatives
  PET MPI Specificity | .762 [.718 to .801]
  SPECT MPI Specificity | .868 [.832 to .898]
Statistical Analysis 1: Comparison: Flurpiridaz F18; Test type: Non-Inferiority or Equivalence — Systematic review of literature and meta-analysis of diagnostic efficacy of SPECT MPI to evaluate the performance criteria of SPECT MPI in studies with various levels of control. Analysis of study protocol number BMS747158-201. Non-inferiority margin (delta) = 7%; p = .945, Z Test — p-Value for specificity comparison of flurpiridaz F18 PET MPI vs. SPECT MPI; one-sided z test for non-inferiority for specificity

10. Secondary Outcome: Overall Summary of Specificity of PET MPI vs SPECT MPI; Image Quality of Excellent or Good
Description: Overall summary of specificity of flurpiridaz F18 PET MPI (qualitative, image quality excellent or good) vs. SPECT MPI by majority rule vs truth standard (angio >/=50% stenosis and confirmed MI). Value represents the number of true negative, i.e. True Negative: Patients with normal MPI and disease negative by the truth standard
Time Frame: 60 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of true negatives
Arm/Group | Flurpiridaz F18 PET MPI
Number analyzed (Participants) | 755
proportion of true negatives
  PET MPI specificity; image quality excellent/good | .769 [.721 to .811]
  SPECT MPI specificity image quality excellent/good | .880 [.841 to .911]
Statistical Analysis 1: Comparison: Flurpiridaz F18 PET MPI; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.954, z Test — p-Value for specificity comparison of flurpiridaz F18 PET MPI vs SPECT MPI for majority rule; image quality excellent/good; p-Value based on on-sided z test for non-inferiority for specificity

11. Secondary Outcome: Image Quality of Rest and Stress (PET vs SPECT).
Description: Overall summary of rest and stress image quality for flurpiridaz F18 PET MPI and SPECT MPI by majority rule. Value represents the number of subject images evaluated as excellent/good and fair/poor
Time Frame: 60 days
Population: as for outcome 1
Measure: Number; unit: percent of images
Arm/Group | Flurpiridaz F18 PET MPI
Number analyzed (Participants) | 755
percent of images
  Rest imaging quality PET MPI; excellent/good | .891
  Rest image quality SPECT MPI; excellent/good | .739
  Stress image quality PET MPI; excellent/good | .976
  Stress image quality SPECT MPI; excellent/good | .869
  Rest image quality PET MPI; fair/poor | .109
  Rest image quality SPECT MPI; fair/poor | .261
  stress image quality PET MPI; fair/poor | .024
  Stress image quality SPECT MPI; fair/poor | .131
Statistical Analysis 1: Comparison: Flurpiridaz F18 PET MPI; Test type: Superiority or Other; p < 0.001, Log Rank

12. Secondary Outcome: Diagnostic Certainty in PET MPI and SPECT MPI
Description: Overall summary of diagnostic certainty in flurpiridaz F18 PET MPI and SPECT MPI by majority rule
Time Frame: 60 days
Population: as for outcome 1
Measure: Number; unit: proportion of patients
Arm/Group | Flurpiridaz F 18
Number analyzed (Participants) | 755
proportion of patients
  PET definitely normal/abnormal | 0.862
  PET probably/equivocal | 0.138
  SPECT definitely normal/abnormal | 0.799
  SPECT probably/equivocal | 0.201
Statistical Analysis 1: Comparison: Flurpiridaz F 18; Test type: Superiority or Other; p < 0.001, McNemar; p-Values are from 2-sided McNemar's test of comparison in proportion of patients with definitely diagnositic certainty between PET and SPECT

ADVERSE EVENTS:
Time Frame: Adverse events occurring from the time of flurpiridaz F 18 rest administration through 14-17 day safety follow up
Description: Affected represents patients with at least one serious adverse event and/or adverse event
Arm/Group | Flurpiridaz F 18
Serious Adverse Events (participants affected / at risk) | 20/795
Other Adverse Events (participants affected / at risk) | 555/795
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flurpiridaz F 18 (N=795)
Angina Pectoris (Cardiac disorders) | 6 (6)
Atrial Flutter (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 2 (2)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1)
Catheter Site Haemorrhage (General disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flurpiridaz F 18 (N=795)
Angina Pectoris (Cardiac disorders) | 119 (119)
Nausea (Gastrointestinal disorders) | 44 (44)
Fatigue (General disorders) | 70 (70)
Non-Cardiac Chest Pain (General disorders) | 58 (58)
Electrocardiogram ST Segment Depressions (Investigations) | 75 (75)
Dizziness (Nervous system disorders) | 43 (43)
Headache (Nervous system disorders) | 129 (129)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 200 (200)
Flushing (Vascular disorders) | 60 (60)
Percutaneous coronary intervention (Surgical and medical procedures) | 72 (72)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less